CLINICAL TRIAL: NCT05385263
Title: Addition of Nivolumab to Standard of Care With Anti-CD-19 CAR-T Cells in Patients With Stable/Progressive DLBCL at Lymphodepletion
Brief Title: Addition of Nivolumab to Anti-CD-19 CAR-T Cells in Patients With Stable/Progressive DLBCL at Lymphodepletion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0804-21
Record Dates: First submitted 2022-04-13; First posted 2022-05-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: All patients enrolled to this study with DLBCL in SD/PD at time of lymphodepletion will be given nivolumab ( 3mg/kg IV) on day +5 Patients with CAR-T expansion<100 cells/microL on day +7 will be given 1 additional dose of nivolumab (3mg/kg IV) on day +19 (two weeks after first dose of nivolumab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIVOLUMAB (Experimental): All patients enrolled will be given nivolumab ( 3mg/kg IV) on day +5 Patients with CAR-T expansion<100 cells/microL on day +7 will be given 1 additional dose of nivolumab (3mg/kg IV) on day +19 (two weeks after first dose of nivolumab).
  Interventions: Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: Nivolumab Injection [Opdivo] — Nivolumab ( 3mg/kg IV) on day +5. If CAR-T expansion<100 cells/microL on day +7 one additional dose of nivolumab (3mg/kg IV) will be given on day +19

SUMMARY:
Progression of DLBCL is the major obstacle for the success of chimeric antigen receptor-T cell (CAR-T) with approximately 60% of the patients relapsing in the first year, and 40% within 3 months, after infusion. While patient with DLBCL in Partial Response/Complete Response at lymphodepletion have a 1-year Progression Free Survival (PFS) of 60-80%, those with Stable Disease/Progressive Disease at time of lymphodepletion have a dismal PFS of 20-30%.

Trials showed that better expansion of CAR-T cells, even in patients with a progressive disease, may overcome this grave prognosis and may result in better PFS

DETAILED DESCRIPTION:
Factors that may introduce resistance to CAR-T. in addition to the bulk of disease, include also expression of check point molecules that eventually interfere with the CAR-T action. The investigator, have recently shown (EBMT 2022, # LWP-03) a real-life data, that day +7 CAR-T concentration in patients with stable or progressive disease (SD/PD) at lymphodepletion segregates patients to those with high CAR-T blood concentrations that achieve a high CR/PR rate after CAR-T infusion ,those with 20-100 CAR-T cells/microL that achieve a lower CR/PR rate after CAR-T infusion, and those with <20 cells/microL that achieve the lowest CR/PR rate after infusion. Thus, the extent of CAR-T cell expansion on day 7 after treatment is a prognostic marker predicting response to treatment in this patient group. Considering all these - patients with SD/PD at time of lymphodepletion, and specifically those with lower CAR-T blood concentrations on day +7 are at a very high risk for early disease progression after CAR-T infusion and, as such, there is an urgent unmet medical need to improve their outcomes.

Addition of anti PD-1 to patients with low expansion of CAR-T cells may overcome the inhibitory effect of PD-1 expression and may result in a better function of the CAR-T and eventually tumor suppression.

Nivolumab is a human monoclonal antibody targeting (programmed death-1 ) PD-1, a negative regulatory molecule expressed by activated T and B lymphocytes. Anti PD-1 treatment has been administered as a single dose or repeated administration in different time points during CAR-T cell therapy. These studies showed that this treatment is safe, well tolerated and does not result in increased CAR-T associated toxicities, mainly cytokine release syndrome(CRS) and immune effector cell associated neurotoxicity(ICANS). The optimal time window to administer these agents for achieving safety and efficacy is not determined.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
2. DLBCL treated with CAR-T targeting CD19 (tisagenlecleucel, axicabtagene ciloleucel, or lisocabtagene maraleucel)
3. PD/SD by PET-CT on the day of lymphodepletion
4. Capable of giving signed informed consent
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. No active CRS or ICANS at time of nivolumab administration

Exclusion Criteria:

1. Hypersensitivity to checkpoints inhibitors
2. CRS grade 3 and above or ICANS any grade on days 0-5 following CAR-T
3. AST (Aspartate transaminase) or ALT (Alanine transaminase) over 3 times the upper limit of normal (ULN) or total bilirubin over 3 times ULN
4. Serum creatinine over 1.5 times ULN or over 1.5 times baseline
5. History of or active autoimmune disease
6. Uncontrolled seizure activity and/or clinically evident progressive encephalopathy
7. Active diarrhea (more than 4 bowel movements per day)
8. Clinically significant uncontrolled illness
9. Active infection requiring antibiotics
10. Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
11. Other active malignancy
12. Females only: Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Overall response at 1 months after CAR-T infusion | One month post CAR-T infusion
  Complete or partial remission rate assessed by PET-CT (Positron Emission Tomography ) at 1 month after combination therapy with nivolumab and CAR-T.

SECONDARY OUTCOMES:
Overall survival at 1 year after CAR-T infusion and nivolumab | One year post CAR-T infusion
  To assess survival of patients at 1 year after infusion of CAR-T and addition of nivolumab.
Duration of response | One year post CAR-T infusion
  Assess duration of disease response after CAR-T infusion
Cytokine release syndrome | One year post CAR-T infusion
  Assesment of cytokine release syndrome according to the American Society for Transplantation and Cellular Therapy (ASTCT) grading system (grade 0-4, 4 being the worse) (TCT. 2019 Apr; 25(4);625-638)
Neurotoxicity | One year post CAR-T infusion
  Assesment of neurotoxicity according to the American Society for Transplantation and Cellular Therapy (ASTCT) grading system (grade 0-4, 4 being the worse) (TCT. 2019 Apr; 25(4);625-638)
Hemophagocytic lymphohistiocytosis (HLH) | One year post CAR-T infusion
  Assesment of HLH according to the Common Terminology Criteria for Adverse Events CTCAE (version 5.0) (grade 3-5, 5 being the worse)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, Prof., Principal Investigator — Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medicak center / BMT Unit, Tel Aviv, Israel

REFERENCES:
- [Derived] Ram R, Amit O, Perry C, Herishanu Y, Avivi I, Sarid N, Apel A, Preis M, Aviv A, Shapira S, Shragai T, Joffe E, Shargian L, Herzog-Tsarfati K, Eylati N, Acria L, Fridberg G, Gold R, Glait-Santar C, Kay S, Gal-Rabinovich K, Rosenberg D, Setter-Marco N, Beyar-Katz O. Addition of Nivolumab Tailored by Expansion of CAR-T Cells in Patients with Stable/Progressive Large B Cell Lymphoma at Lymphodepletion-A Phase 2, Prospective Interventional Study. Transplant Cell Ther. 2024 Dec;30(12):1178-1188. doi: 10.1016/j.jtct.2024.09.024. Epub 2024 Oct 11. PMID 39396632